CLINICAL TRIAL: NCT03320486
Title: Phase 3, Multicenter, Double-blind, Randomized, Non-inferiority Clinical Trial of Dapaconazole Cream 2% (Biolab Sanus Farmacêutica Ltda.) Versus Ketoconazole Cream 2% (Nizoral®, Janssen-Cilag Farmacêutica Ltda.) in Patients With Tinea Pedis
Brief Title: Non-inferiority Trial of Dapaconazole Versus Ketoconazole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDN 018/16
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Tinea Pedis
Keywords: Mycoses; Dermatomycoses; Antifugal Agents; Dapaconazole
MeSH Terms: conditions — Tinea Pedis; Mycoses; Dermatomycoses | interventions — 1-(2-(2,4-dichlorophenyl)-2-(4-(trifluoromethyl)benzyloxy)ethyl)-1H-imidazole; Ketoconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - dapaconazole cream 2% (Experimental): Topical application of dapaconazole cream 2%, once daily, during 42 days.
  Interventions: Drug: Dapaconazole
- Group 2 - ketoconazole cream 2% (Active Comparator): Topical application of ketoconazole cream 2%, once daily, during 42 days.
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Dapaconazole — Application of 1 to 3 grams, depending on the lesion extension, per affected foot.
  Other Names: Zilt
  Arms: Group 1 - dapaconazole cream 2%
Drug: Ketoconazole — Application of 1 to 3 grams, depending on the lesion extension, per affected foot.
  Other Names: Nizoral®
  Arms: Group 2 - ketoconazole cream 2%

SUMMARY:
The main purpose of this study is to demonstrate that dapaconazole cream 2% (experimental drug) is non-inferior to ketoconazole cream 2% (Nizoral® - active comparator) for the treatment of dermatological lesions of Tinea pedis, when applied to the skin (topically) once daily during 28 days. Additionally, the safety and tolerability aspects will be evaluated in a descriptive way, through the observation of the incidence of adverse events.

DETAILED DESCRIPTION:
This is a non-inferiority, phase 3, multicenter, double-blind, randomized (allocation of treatment), balanced, controlled (active comparator) trial, with two parallel groups in a 1:1 proportion.

Randomization will depend on inclusion/exclusion criteria, taking into account the confirmation of diagnosis by the direct mycological test performed during the screening phase. However, cases whose diagnosis is not additionally confirmed by positive fungal culture (sampled during the screening phase) will be excluded from the efficacy analysis.

Participants will show up to the clinic, for treatment, during 42 consecutive days, when one of the investigational products (according to the randomization) will be applied by a blind member of the study staff. A non-blind member of the study staff will weigh the corresponding investigational product and pass on to the blind member only a spatula with the weighed product, in order to maintain the blinded aspect of the trial.

For exploratory purposes, clinical and mycological evaluations will also be performed after 7 and after 14 days of treatment.

Safety analysis will be performed considering all the randomized patients to which at least one dose of the investigational products has been applied, regardless of the result of the fungal culture.

Conclusion of non-inferiority will be based on the per protocol set. It will be deemed as per protocol those participants who do not miss more than 20% of the applications and, also, no more than four consecutive application days.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged from 18 to 65 years old, male, or female with no childbearing potential or who are using an effective contraceptive method and who do not plan to become pregnant during the study period.
* Presence of dermatological lesion(s) of Tinea pedis, with a global clinical severity score ≥ 4, being a minimum score of 2 for itching or desquamation/maceration and a minimum score of 2 for erythema, having, also, the diagnosis confirmed by direct mycological (KOH) test.
* No previous treatment with antimycotic medication, in the last 2 months, for the current dermatologic lesion.
* No evidence of other significant diseases, that, at the investigator's discretion, may affect the participation in the clinical trial, in accordance with the protocol requirements.
* Ability to understand the nature and the objective of the clinical trial, including the risks and possible side effects; intention to cooperate with the investigator and act in accordance with the protocol requirements, as confirmed by the informed consent form signature.

Exclusion Criteria:

* Existing hepatic and/or renal diseases or other pathologic findings, which might interfere with the safety and tolerability of the active ingredients.
* Screening laboratory tests presenting deviations deemed as clinically significant, which, due to possible risks, prevents the participation in clinical trial.
* Known hypersensitivity to ketoconazole or to chemically related compounds (azoles) or to the compounds of the investigational products.
* Participants with severe or multiple drugs allergies, unless judged by the investigator as not clinically relevant to the participation in the clinical trial.
* Positive anti human immunodeficiency virus (anti-HIV) test, positive Hepatitis B Surface Antigen (HBs-Ag) test or positive anti hepatitis C virus (anti-HCV) test.
* Treatment, within 3 months prior to the start of the clinical trial treatment, with any drug known to have a well-established toxic potential to major organs.
* Pregnant or lactating women
* Participation in any clinical trial, or intake of any investigational product, within the last twelve months prior to the inclusion in the clinical trial.
* Presence of onychomycosis.
* Presence of "Moccasin type" Tinea pedis.
* Presence of infected Tinea pedis, or any other infection or pathology that may confuse the treatment evaluation.
* History of drug addiction.
* Diseases that may alter the immune system and, consequently, the host's response to the fungal presence (immunosuppressed participants), as well as the use of systemic immunosuppressive drugs, chemotherapy or radiotherapy, during the 3 months prior to the start of treatment.
* Use of drugs that may interfere with the assessment of the results, as well as use of topical immunosuppressants, topical antibiotics or topical corticosteroids, within 2 months prior to the start of treatment.
* Use of antipruriginous drugs, including antihistaminics, within 72 hours prior to the start of treatment.
* History of alcohol dependence and/or regular intake of alcoholic food or beverages containing ≥ 20 g of pure ethanol per day.
* Any prior treatment for the present lesion which, at investigator discretion, may interfere with the objectives of the clinical trial.
* Participants who might be non-compliant to the study treatment and/or to the requirements and procedures of the protocol.
* Participants who are unable to understand written and verbal instructions, in particular those regarding the risks and inconveniences to which they will be exposed during the participation in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with therapeutic cure | 28 days of treatment
  Proportion of participants, in each treatment group, who achieved therapeutic cure, defined as both clinical cure and mycological cure, on the assessment performed after 28 days of treatment.
  Clinical cure is defined as a score ≤ 2 for the sum of scores attributed to each sign or symptom (erythema, maceration/peeling, fissuring/cracking, itching and burning) as evaluated by a four-point categorical scale (0=absent, 1=mild, 2=moderate, 3=severe).
  Mycological cure is defined as negative result for the direct mycological examination (potassium hydroxide [KOH] test) and a negative fungal culture.

SECONDARY OUTCOMES:
Proportion of participants with therapeutic cure | 42 days of treatment
  Proportion of participants, in each treatment group, who achieved therapeutic cure, on the assessment performed after 42 days of treatment.
Proportion of participants maintaining therapeutic cure | 14 (±3) days after the end of treatment
  Proportion of participants, in each treatment group, maintaining the therapeutic cure in the evaluation performed approximately 14 days after the end of the 42 days treatment period.
Proportion of participants maintaining therapeutic cure | 28 (±5) days after the end of treatment
  Proportion of participants, in each treatment group, maintaining the therapeutic cure in the evaluation performed approximately 28 days after the end of the 42 days treatment period.
Number of days until clinical cure | up to 42 days
  Number of days elapsed between the day of start of treatment and the day when the clinical cure is diagnosed, according to the daily assessment, in each treatment group.
Number of adverse events per participant | up to 80 (±5) days
  Number of adverse events, in each treatment group, including clinically relevant alterations of vital signs and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto De Nucci, MD, Principal Investigator — Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME
Locations (1):
- Galeno Desenvolvimento de Pesquisas Clinicas Ltda. - ME, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No